CLINICAL TRIAL: NCT05887401
Title: A Pilot Randomized Factorial Trial to Promote Physical Activity and Healthy Eating Among Young Adult Cancer Survivors
Brief Title: Physical Activity and Healthy Eating Among Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: LCCC2233; T32CA057726 (NIH)
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Physical Activity; Neoplasms; Cancer
MeSH Terms: conditions — Motor Activity; Neoplasms | interventions — Green Or; Dyrk Kinases; YES1 protein, human

STUDY DESIGN:
Intervention Model Description: This study uses a full factorial experimental design testing the efficacy of four intervention components, each with two levels
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Green Foods Monitoring, Daily Nutrition Goals, Supportive Text Messages, All Lessons Once (Experimental): Core + Green Foods Monitoring + Nutrition Goals + Supportive Text Messages + Lessons Weekly
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Green); Behavioral: Nutrition Goals (Yes); Behavioral: Supportive Text Messages (Yes); Behavioral: Lesson Delivery (Once)
- Green Foods Monitoring, Daily Nutrition Goals, Supportive Text Messages, Weekly Lessons (Experimental): Core + Green Foods Monitoring + Nutrition Goals + Supportive Text Messages + Weekly Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Green); Behavioral: Nutrition Goals (Yes); Behavioral: Supportive Text Messages (Yes); Behavioral: Lesson Delivery (Weekly)
- Green Foods Monitoring, Daily Nutrition Goals, No Text Messages, All Lessons Once (Experimental): Core + Green Foods Monitoring + Nutrition Goals + No Supportive Text Messages + All Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Green); Behavioral: Nutrition Goals (Yes); Behavioral: Supportive Text Messages (No); Behavioral: Lesson Delivery (Once)
- Green Foods Monitoring, Daily Nutrition Goals, No Supportive Text Messages, Weekly Lessons (Experimental): Core + Green Foods Monitoring + Nutrition Goals + No Supportive Text Messages + Weekly Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Green); Behavioral: Nutrition Goals (Yes); Behavioral: Supportive Text Messages (No); Behavioral: Lesson Delivery (Weekly)
- Green Foods Monitoring, No Nutrition Goals, Supportive Text Messages, All Lessons Once (Experimental): Core + Green Foods Monitoring + No Nutrition Goals + Supportive Text Messages + All Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Green); Behavioral: Nutrition Goals (No); Behavioral: Supportive Text Messages (Yes); Behavioral: Lesson Delivery (Once)
- Green Foods Monitoring, No Nutrition Goals, Supportive Text Messages, Weekly Lessons (Experimental): Core + Green Foods Monitoring + No Nutrition Goals + Supportive Text Messages + Weekly Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Green); Behavioral: Nutrition Goals (No); Behavioral: Supportive Text Messages (Yes); Behavioral: Lesson Delivery (Weekly)
- Green Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, All Lessons Once (Experimental): Core + Green Foods Monitoring + No Nutrition Goals + No Supportive Text Messages + All Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Green); Behavioral: Nutrition Goals (No); Behavioral: Supportive Text Messages (No); Behavioral: Lesson Delivery (Once)
- Green Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, Weekly Lessons (Experimental): Core + Green Foods Monitoring + No Nutrition Goals + No Supportive Text Messages + Weekly Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Green); Behavioral: Nutrition Goals (No); Behavioral: Supportive Text Messages (No); Behavioral: Lesson Delivery (Weekly)
- Red Foods Monitoring, Nutrition Goals, Supportive Text Messages, All Lessons Once (Experimental): Core + Red Foods Monitoring + Nutrition Goals + Supportive Text Messages + All Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Red); Behavioral: Nutrition Goals (Yes); Behavioral: Supportive Text Messages (Yes); Behavioral: Lesson Delivery (Once)
- Red Foods Monitoring, Nutrition Goals, Supportive Text Messages, Weekly Lessons (Experimental): Core + Red Foods Monitoring + Nutrition Goals + Supportive Text Messages + Weekly Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Red); Behavioral: Nutrition Goals (Yes); Behavioral: Supportive Text Messages (Yes); Behavioral: Lesson Delivery (Weekly)
- Red Foods Monitoring, Nutrition Goals, No Supportive Text Messages, All Lessons Once (Experimental): Core + Red Foods Monitoring + Nutrition Goals + No Supportive Text Messages + All Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Red); Behavioral: Nutrition Goals (Yes); Behavioral: Supportive Text Messages (No); Behavioral: Lesson Delivery (Once)
- Red Foods Monitoring, Nutrition Goals, No Supportive Text Messages, Weekly Lessons (Experimental): Core + Red Foods Monitoring + Nutrition Goals + No Supportive Text Messages + Weekly Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Red); Behavioral: Nutrition Goals (Yes); Behavioral: Supportive Text Messages (No); Behavioral: Lesson Delivery (Weekly)
- Red Foods Monitoring, No Nutrition Goals, Supportive Text Messages, All Lessons Once (Experimental): Core + Red Foods Monitoring + No Nutrition Goals + Supportive Text Messages + All Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Red); Behavioral: Nutrition Goals (No); Behavioral: Supportive Text Messages (Yes); Behavioral: Lesson Delivery (Once)
- Red Foods Monitoring, No Nutrition Goals, Supportive Text Messages, Weekly Lessons (Experimental): Core + Red Foods Monitoring + No Nutrition Goals + Supportive Text Messages + Weekly Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Red); Behavioral: Nutrition Goals (No); Behavioral: Supportive Text Messages (Yes); Behavioral: Lesson Delivery (Weekly)
- Red Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, All Lessons Once (Experimental): Core + Red Foods Monitoring + No Nutrition Goals + No Supportive Text Messages + All Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Red); Behavioral: Nutrition Goals (No); Behavioral: Supportive Text Messages (No); Behavioral: Lesson Delivery (Once)
- Red Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, Weekly Lessons (Experimental): Core + Red Foods Monitoring + No Nutrition Goals + No Supportive Text Messages + Weekly Lessons
  Interventions: Behavioral: Core Intervention; Behavioral: Simplified Dietary Monitoring (Red); Behavioral: Nutrition Goals (No); Behavioral: Supportive Text Messages (No); Behavioral: Lesson Delivery (Weekly)

INTERVENTIONS:
Behavioral: Core Intervention — The core intervention will include behavioral lessons, activity tracker, weekly adaptive physical activity goals, weekly tailored feedback summary.
Behavioral: Simplified Dietary Monitoring (Green) — Simplified diet monitoring using smartphone tracking of green foods using a traffic light approach.
  Arms: Green Foods Monitoring, Daily Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Green Foods Monitoring, Daily Nutrition Goals, No Text Messages, All Lessons Once; Green Foods Monitoring, Daily Nutrition Goals, Supportive Text Messages, All Lessons Once; Green Foods Monitoring, Daily Nutrition Goals, Supportive Text Messages, Weekly Lessons; Green Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, All Lessons Once; Green Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Green Foods Monitoring, No Nutrition Goals, Supportive Text Messages, All Lessons Once; Green Foods Monitoring, No Nutrition Goals, Supportive Text Messages, Weekly Lessons
Behavioral: Simplified Dietary Monitoring (Red) — Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Arms: Red Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, All Lessons Once; Red Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, No Nutrition Goals, Supportive Text Messages, All Lessons Once; Red Foods Monitoring, No Nutrition Goals, Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, Nutrition Goals, No Supportive Text Messages, All Lessons Once; Red Foods Monitoring, Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, Nutrition Goals, Supportive Text Messages, All Lessons Once; Red Foods Monitoring, Nutrition Goals, Supportive Text Messages, Weekly Lessons
Behavioral: Nutrition Goals (Yes) — Participant will be assigned a personalized weekly nutrition goal related to nutrition monitoring condition.
  Arms: Green Foods Monitoring, Daily Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Green Foods Monitoring, Daily Nutrition Goals, No Text Messages, All Lessons Once; Green Foods Monitoring, Daily Nutrition Goals, Supportive Text Messages, All Lessons Once; Green Foods Monitoring, Daily Nutrition Goals, Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, Nutrition Goals, No Supportive Text Messages, All Lessons Once; Red Foods Monitoring, Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, Nutrition Goals, Supportive Text Messages, All Lessons Once; Red Foods Monitoring, Nutrition Goals, Supportive Text Messages, Weekly Lessons
Behavioral: Nutrition Goals (No) — Participant will not be assigned a personalized weekly nutrition goal.
  Arms: Green Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, All Lessons Once; Green Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Green Foods Monitoring, No Nutrition Goals, Supportive Text Messages, All Lessons Once; Green Foods Monitoring, No Nutrition Goals, Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, All Lessons Once; Red Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, No Nutrition Goals, Supportive Text Messages, All Lessons Once; Red Foods Monitoring, No Nutrition Goals, Supportive Text Messages, Weekly Lessons
Behavioral: Supportive Text Messages (Yes) — Participant will receive up to 5 supportive text-messages from the study staff per week.
  Arms: Green Foods Monitoring, Daily Nutrition Goals, Supportive Text Messages, All Lessons Once; Green Foods Monitoring, Daily Nutrition Goals, Supportive Text Messages, Weekly Lessons; Green Foods Monitoring, No Nutrition Goals, Supportive Text Messages, All Lessons Once; Green Foods Monitoring, No Nutrition Goals, Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, No Nutrition Goals, Supportive Text Messages, All Lessons Once; Red Foods Monitoring, No Nutrition Goals, Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, Nutrition Goals, Supportive Text Messages, All Lessons Once; Red Foods Monitoring, Nutrition Goals, Supportive Text Messages, Weekly Lessons
Behavioral: Supportive Text Messages (No) — Participant will not receive supportive text-messages.
  Arms: Green Foods Monitoring, Daily Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Green Foods Monitoring, Daily Nutrition Goals, No Text Messages, All Lessons Once; Green Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, All Lessons Once; Green Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, All Lessons Once; Red Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, Nutrition Goals, No Supportive Text Messages, All Lessons Once; Red Foods Monitoring, Nutrition Goals, No Supportive Text Messages, Weekly Lessons
Behavioral: Lesson Delivery (Once) — All behavioral lessons will be made available to participant simultaneously.
  Arms: Green Foods Monitoring, Daily Nutrition Goals, No Text Messages, All Lessons Once; Green Foods Monitoring, Daily Nutrition Goals, Supportive Text Messages, All Lessons Once; Green Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, All Lessons Once; Green Foods Monitoring, No Nutrition Goals, Supportive Text Messages, All Lessons Once; Red Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, All Lessons Once; Red Foods Monitoring, No Nutrition Goals, Supportive Text Messages, All Lessons Once; Red Foods Monitoring, Nutrition Goals, No Supportive Text Messages, All Lessons Once; Red Foods Monitoring, Nutrition Goals, Supportive Text Messages, All Lessons Once
Behavioral: Lesson Delivery (Weekly) — A new behavioral lesson will be made available to participant weekly throughout the 12 weeks.
  Arms: Green Foods Monitoring, Daily Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Green Foods Monitoring, Daily Nutrition Goals, Supportive Text Messages, Weekly Lessons; Green Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Green Foods Monitoring, No Nutrition Goals, Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, No Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, No Nutrition Goals, Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, Nutrition Goals, No Supportive Text Messages, Weekly Lessons; Red Foods Monitoring, Nutrition Goals, Supportive Text Messages, Weekly Lessons

SUMMARY:
The purpose of this pilot randomized factorial trial is to test the feasibility, acceptability, and effects of a theory-based mobile physical activity and nutrition intervention designed specifically for young adult cancer survivors to increase physical activity and diet quality.

DETAILED DESCRIPTION:
There are around 1 million young adult cancer survivors in the United States. Young adult cancer survivors are an underserved and vulnerable subgroup of survivors that experience increased risk for chronic health conditions like cardiovascular disease, metabolic syndrome, secondary cancers, premature aging, and premature death. Modifiable lifestyle factors contribute to and compound risks for late and long-term health effects from cancer and its treatment, making them high-impact targets for behavioral interventions. International consensus guidelines recommend cancer survivors of all ages be physically active, consume a healthy diet, and achieve and maintain a healthy weight. Fewer than half of young adult cancer survivors meet guideline recommendations for vegetable intake, physical activity and the majority self-report having an overweight/obese BMI. To date, there are few physical activity interventions, and no nutritional interventions designed specifically for young adult cancer survivors. Digital behavior change interventions have emerged as feasible and efficacious approaches to reach and address unmet needs among young adult cancer survivors as they overcome barriers of time, flexibility, affordability, and access. Reaching these populations has been facilitated by digital tools like wearable devices that enable real-time data capture to guide the provision of individualized feedback and tailored goal setting based on personal progress. This pilot trial will use the Multiphase Optimization Strategy (MOST), an engineering-inspired framework, and a highly efficient experimental design to evaluate the feasibility of 4 intervention components to improve physical activity and nutrition behaviors among young adult cancer survivors. Young adult cancer survivors (n=80), diagnosed between ages 18-39, will be recruited to receive a core 3-month digital physical activity and nutrition intervention that includes evidence-based lessons and behavioral skills training with an emphasis on adherence to American Cancer Society (ACS) guidelines for cancer survivors and self-monitoring of physical activity and dietary behaviors. Additionally, participants will be randomized to four intervention components--each with two levels-- including: 1) simplified dietary tracking (daily tracking of green (low-calorie, high nutrients) vs. red (high-calorie, high-fat, low nutrients) foods), 2) dietary goals using simplified approach (daily goals vs. no goals), 3) supportive text messages (yes vs. no), 4) lesson delivery (all provided once vs. weekly). Assessments of outcomes will be conducted at baseline, 6 weeks, and 3 months to accomplish the following specific aims: 1) Evaluate the feasibility and acceptability the intervention at 3 months; 2) Evaluate intervention effects on change in physical activity and diet quality; 3) Evaluate intervention effects on secondary outcomes at 6 weeks and 3 months; and 4) Explore whether theoretical constructs (perceived competence, self-regulation, self-efficacy, and perceived relatedness) mediated the effects of the intervention on change in health behaviors at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Current age 18-39 years at the time of consent
* Diagnosed with invasive cancer malignancy between the ages of 15-39 years
* Diagnosed with invasive malignancy in the last 10 years of diagnosis, and with no evidence of progressive disease or second primary cancers
* Completed active cancer directed therapy (cytotoxic chemotherapy, radiation therapy and/or definitive surgical intervention), except may be receiving "maintenance" therapy to prevent recurrences
* No pre-existing medical conditions(s) that preclude adherence to an unsupervised exercise program including cardiovascular disease, congestive heart failure, pulmonary conditions, renal disease, and severe orthopedic conditions
* Not currently meeting guideline recommendations of 150 minutes/week moderate to vigorous physical activity (self-report) and guideline recommendations for fruit and vegetable consumption (self-report)
* Have the ability to read, write and speak English
* Have access to the Internet on at least a weekly basis
* Possession and usage of an Internet e-mail address or willingness to sign up for a free email account (e.g., gmail)
* Have smartphone with internet access and text messaging plan
* Be willing to be randomized to any condition

Exclusion Criteria:

* History of heart attack or stroke within past 6 months
* Untreated hypertension, hyperlipidemia, or diabetes, unless permission is provided by their health care provider
* Health problems which preclude ability to walk for physical activity
* Report a diagnosis of psychiatric diseases (schizophrenia, bipolar disorder, depression leading to hospitalization in the past year), drug or alcohol dependency
* Report a past diagnosis of or treatment for a Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) eating disorder (anorexia nervosa or bulimia nervosa)
* Plans for major surgery (e.g., breast reconstruction) during the study time frame
* Current participation in another physical activity or weight control program
* Currently using prescription weight loss medications
* Currently pregnant, pregnant within the past 6 months, or planning to become pregnant within the next 6 months
* Currently exercising > 150 minutes/week of moderate-to-vigorous intensity physical activity
* Currently consuming > 5 servings of fruits and vegetables/day.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin M Coffman, MA, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from October 2023 and April 2024; remote recruitment across the continental United States. 220 individuals completed the online screening survey; 83 were initially eligible; out of those, 11 completed informed consent but were ineligible due to no longer being interested in participating or incomplete baseline measurement procedures, and 72 completed informed consent and all baseline assessment procedures and were randomized and enrolled in the study.
Pre-assignment Details: Individuals who signed informed consent and then completed all baseline measurement procedures (online surveys and remote weight measurements) and remained eligible were considered enrolled and were randomized to 1 of 16 conditions.
Groups:
- Condition 1: Core + Green Foods Monitoring + Nutrition Goals + Supportive Text Messages + All Lessons
- Condition 2: Core + Green Foods Monitoring + Nutrition Goals + Supportive Text Messages + Weekly Lessons
- Condition 3: Core + Green Foods Monitoring + Nutrition Goals + No Supportive Text Messages + All Lessons
- Condition 4: Core + Green Foods Monitoring + Nutrition Goals + No Supportive Text Messages + Weekly Lessons
- Condition 5: Core + Green Foods Monitoring + No Nutrition Goals + Supportive Text Messages + All Lessons
- Condition 6: Core + Green Foods Monitoring + No Nutrition Goals + Supportive Text Messages + Weekly Lessons
- Condition 7: Core + Green Foods Monitoring + No Nutrition Goals + No Supportive Text Messages + All Lessons
- Condition 8: Core + Green Foods Monitoring + No Nutrition Goals + No Supportive Text Messages + Weekly Lessons
- Condition 9: Core + Red Foods Monitoring + Nutrition Goals + Supportive Text Messages + All Lessons
- Condition 10: Core + Red Foods Monitoring + Nutrition Goals + Supportive Text Messages + Weekly Lessons
- Condition 11: Core + Red Foods Monitoring + Nutrition Goals + No Supportive Text Messages + All Lessons
- Condition 12: Core + Red Foods Monitoring + Nutrition Goals + No Supportive Text Messages + Weekly Lessons
- Condition 13: Core + Red Foods Monitoring + No Nutrition Goals + Supportive Text Messages + All Lessons
- Condition 14: Core + Red Foods Monitoring + No Nutrition Goals + Supportive Text Messages + Weekly Lessons
- Condition 15: Core + Red Foods Monitoring + No Nutrition Goals + No Supportive Text Messages + All Lessons
- Condition 16: Core + Red Foods Monitoring + No Nutrition Goals + No Supportive Text Messages + Weekly Lessons
Period: Overall Study
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16
Started | 4 | 5 | 4 | 4 | 3 | 4 | 6 | 4 | 2 | 5 | 5 | 5 | 6 | 7 | 4 | 4
Completed | 4 | 4 | 3 | 2 | 3 | 4 | 6 | 4 | 1 | 3 | 3 | 4 | 6 | 7 | 4 | 3
Not Completed | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants, N=72.
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16 | Total
Number analyzed (Participants) | 4 | 5 | 4 | 4 | 3 | 4 | 6 | 4 | 2 | 5 | 5 | 5 | 6 | 7 | 4 | 4 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (1.81) | 34.1 (6.15) | 29.2 (7.36) | 31.2 (8.13) | 38.6 (1.18) | 34.5 (8.07) | 34.8 (3.14) | 34.1 (5.77) | 34.2 (0.92) | 35.2 (4.03) | 31.6 (7.06) | 31.8 (5.34) | 32.2 (5.48) | 36.6 (2.82) | 29.4 (5.56) | 33.5 (3.45) | 33.5 (5.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 4 | 4 | 4 | 3 | 2 | 4 | 5 | 3 | 2 | 4 | 5 | 4 | 5 | 5 | 4 | 4 | 62
  Sex: Male | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  White | 3 | 3 | 3 | 3 | 3 | 4 | 5 | 3 | 2 | 4 | 5 | 5 | 4 | 6 | 3 | 4 | 60
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 13
  Not Hispanic or Latino | 4 | 1 | 3 | 3 | 3 | 3 | 4 | 3 | 2 | 2 | 5 | 5 | 5 | 7 | 3 | 4 | 57
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: Participants]
  United States | 4 | 5 | 4 | 4 | 3 | 4 | 6 | 4 | 2 | 5 | 5 | 5 | 6 | 7 | 4 | 4 | 72
Weight (lb) [Mean (Standard Deviation); unit: pounds] — Weight was objectively measured at the participant's home. Participants were instructed to weigh themselves first thing in the morning, in light clothing, without shoes, at each assessment time point. Participants entered their weight in the study app and uploaded a picture of their feet on the scale with the number visible for verification.
  pounds | 163.50 (24.61) | 179.20 (60.40) | 136.25 (18.08) | 168.00 (36.12) | 167.33 (8.96) | 174.00 (8.04) | 188.33 (26.27) | 182.00 (85.12) | 203.50 (72.83) | 169.60 (48.28) | 175.80 (50.31) | 182.60 (63.87) | 183.17 (26.07) | 180.14 (31.39) | 156.25 (39.02) | 173.75 (28.48) | 174.31 (40.51)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.04 (6.88) | 29.30 (9.29) | 21.66 (2.78) | 26.22 (6.37) | 26.83 (1.90) | 29.72 (2.57) | 33.01 (8.74) | 34.84 (21.55) | 32.33 (15.22) | 25.20 (6.67) | 30.49 (8.37) | 27.24 (6.52) | 30.24 (4.22) | 28.13 (4.06) | 26.82 (7.47) | 26.31 (6.11) | 28.46 (7.92)
Physical Activity (MVPA) [Mean (Standard Deviation); unit: min/wk] — Objective moderate-to-vigorous physical activity (MVPA) measured via Fitbit
  min/wk | 173.25 (37.69) | 176.80 (247.80) | 73.25 (63.89) | 91.75 (52.00) | 395.67 (143.83) | 184.00 (258.98) | 250.00 (218.85) | 200.25 (150.93) | 50.50 (2.12) | 280.00 (195.54) | 124.00 (200.22) | 152.00 (106.84) | 122.50 (104.09) | 203.14 (188.81) | 177.75 (101.74) | 221.00 (27.29) | 181.86 (161.93)
Diet [Mean (Standard Deviation); unit: Points] — Baseline Health Eating Index (HEI) score. HEI consists of 13 component scores, including: total fruit, whole fruit, total protein foods, total vegetables, greens and beans, whole grains, dairy, seafood and plant proteins, fatty acids, sodium, refined grains, added sugars, and saturated fats. The summation of the 13 component scores ranges from 0 to 100, with higher scores indicating closer compliance with the Dietary Guidelines for Americans
  Points | 46.55 (15.21) | 56.52 (18.52) | 39.52 (9.13) | 57.93 (12.33) | 64.93 (3.81) | 46.93 (10.16) | 51.51 (14.45) | 54.26 (12.95) | 66.39 (14.12) | 57.53 (9.58) | 49.33 (12.88) | 54.51 (14.79) | 53.97 (11.88) | 53.34 (9.96) | 50.02 (7.69) | 48.30 (15.05) | 52.74 (12.58)

OUTCOME MEASURES:

1. Primary Outcome: Accrual Rate
Description: Number of participants who agreed to participate divided by the number of months of recruitment.
Time Frame: End of study enrollment period (7 months).
Population: Because this measure pertains to the study as a whole, the number of participants is not reported by arm.
Measure: Number; unit: Participants per month
Groups:
- Participants Recruited: All eligible participants who agreed to participate in the intervention.
Arm/Group | Participants Recruited
Number analyzed (Participants) | 83
Participants per month | 12

2. Primary Outcome: Participation Rate
Description: Percentage of consented participants who were randomized.
Time Frame: End of study enrollment period (7 months).
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Recruited
Number analyzed (Participants) | 83
Participants | 72

3. Primary Outcome: Retention Rate
Description: Number of intervention participants who completed 3-month measures divided by the number randomized to intervention arms.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16
Number analyzed (Participants) | 4 | 5 | 4 | 4 | 3 | 4 | 6 | 4 | 2 | 5 | 5 | 5 | 6 | 7 | 4 | 4
Participants | 4 | 4 | 3 | 2 | 3 | 4 | 6 | 4 | 1 | 3 | 3 | 4 | 6 | 7 | 4 | 3

4. Secondary Outcome: Acceptability: How Satisfied Are You Overall With the Program You Received?
Description: 1-item measure; a benchmark of 80% of participants answering "somewhat" or "very" satisfied would indicate acceptability
Time Frame: 3 months
Population: Among completers of the 12-week questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- Nutrition Goals (Yes): Participants will be assigned a personalized weekly nutrition goal related to the nutrition monitoring condition.
- Nutrition Goals (No): Participants will not be assigned a personalized weekly nutrition goal.
- Supportive Text Messages (Yes): Participants will receive up to 5 supportive text messages from the study staff per week.
- Supportive Text Messages (No): Participants will not receive supportive text messages.
- Lesson Delivery (Once): All behavioral lessons will be made available to participants simultaneously at the beginning of the intervention.
- Lesson Delivery (Weekly): A new behavioral lesson will be made available to participants weekly throughout the 12 weeks.
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly)
Number analyzed (Participants) | 30 | 30 | 24 | 36 | 31 | 29 | 30 | 30
Participants | 24 | 27 | 20 | 31 | 26 | 25 | 25 | 26

5. Secondary Outcome: Adherence to Physical Activity Monitoring.
Description: Number of days physical activity tracked, as measured by Fitbit.
Time Frame: Through study completion, 3 months.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly)
Number analyzed (Participants) | 34 | 38 | 34 | 38 | 36 | 36 | 34 | 38
Days | 81.5 (21.0) [65.8 to 84] | 70.8 (21.0) [66.5 to 83] | 79 (25.1) [51 to 83] | 83 [77.2 to 84] | 83 [73.2 to 84] | 79 [58.8 to 83.2] | 81.5 [76 to 83] | 83 [60 to 84]

6. Secondary Outcome: Adherence to Diet Self-monitoring
Description: Number of days of complete dietary tracking.
Time Frame: Through study completion, 3 months.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly)
Number analyzed (Participants) | 34 | 38 | 34 | 38 | 36 | 36 | 34 | 38
Days | 43 [19.5 to 60] | 49.5 [17 to 61.5] | 39.5 [9 to 60] | 52 [27.2 to 59.8] | 52 [27 to 69.2] | 35 [8.5 to 57] | 48.5 [27 to 60] | 44.5 [6.75 to 60]

7. Secondary Outcome: Moderate-to-vigorous Physical Activity (Objective)
Description: Estimated mean change in MVPA from baseline to 3 months for each of the two levels of each component obtained from intent-to-treat (ITT) linear mixed models of analysis of variance.
Time Frame: Baseline, 3 months.
Population: ITT: all randomized participants using all available MVPA data.
Measure: Mean (95% Confidence Interval); unit: min/wk
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly)
Number analyzed (Participants) | 34 | 38 | 34 | 38 | 36 | 36 | 34 | 38
min/wk | 52.78 [-36.06 to 141.62] | 70.12 [-16.10 to 156.33] | 69.70 [-24.96 to 164.35] | 53.20 [-28.21 to 134.61] | 75.94 [-13.61 to 165.48] | 46.96 [-40.23 to 134.16] | 69.23 [-20.61 to 159.06] | 53.67 [-33.31 to 140.65]
Statistical Analysis 1: Comparison: Simplified Dietary Monitoring (Green) vs Simplified Dietary Monitoring (Red) vs Nutrition Goals (Yes) vs Nutrition Goals (No) vs Supportive Text Messages (Yes) vs Supportive Text Messages (No) vs Lesson Delivery (Once) vs Lesson Delivery (Weekly); Test type: Superiority — ITT analysis using linear mixed models comparing MVPA change over time (from baseline to 3 months). We fit a linear mixed model that included a random effect for participant and predictors (fixed effects) included time (baseline vs. follow-up) and all 4 factors; p = 0.02, Mixed Models Analysis — The reported p-value reflects the change across time for the full sample; DF(2, 119); Mean Difference (Net) = 61.45, 95% CI 2-sided [9.95 to 112.95] — The positive parameter estimate indicates an increase in MVPA over time for the full sample
Statistical Analysis 2: Comparison: Simplified Dietary Monitoring (Green) vs Simplified Dietary Monitoring (Red); ITT analysis for factor 1 (dietary self-monitoring) using linear mixed models comparing the effect of simplified dietary monitoring (green vs. red) on MVPA change over time (from baseline to 3 months); Test type: Superiority; p = 0.65, Mixed Models Analysis; DF(1, 69); Mean Difference (Net) = 21.36, 95% CI 2-sided [-70.89 to 113.61] — Green food monitoring (reference) vs red food monitoring; a positive estimation parameter indicates that the reference group had greater increases in MVPA over time
Statistical Analysis 3: Comparison: Nutrition Goals (Yes) vs Nutrition Goals (No); ITT analysis for factor 2 (dietary goals) using linear mixed models comparing the effect of dietary goals (yes vs. no) on MVPA change over time (from baseline to 3 months); Test type: Superiority; p = 0.20, Mixed Models Analysis; DF(1,70); Mean Difference (Net) = -60.05, 95% CI 2-sided [-152.40 to 32.39] — Nutrition goals (yes; reference) vs no goals provided; a negative estimation parameter indicates that the non-referent group had greater increases in MVPA over time
Statistical Analysis 4: Comparison: Supportive Text Messages (Yes) vs Supportive Text Messages (No); ITT analysis for factor 3 (supportive text messages) using linear mixed models comparing the effect of text messages (yes vs. no) on MVPA change over time (from baseline to 3 months); Test type: Superiority; p = 0.53, Mixed Models Analysis; DF(1,70); Mean Difference (Net) = 29.52, 95% CI 2-sided [-63.07 to 122.11] — Supportive text messages (yes; reference) vs no text messages; a positive estimation parameter indicates that the reference group had greater increases in MVPA over time
Statistical Analysis 5: Comparison: Lesson Delivery (Once) vs Lesson Delivery (Weekly); ITT analysis for factor 4 (lesson delivery) using linear mixed models comparing the effect of lesson timing (once vs. weekly) on MVPA change over time (from baseline to 3 months); Test type: Superiority; p = 0.66, Mixed Models Analysis; DF(1,70); Mean Difference (Final Values) = -20.5, 95% CI 2-sided [-113.26 to 72.27] — Lesson delivery once (reference) vs weekly; a negative estimation parameter indicates that the non-referent group had greater increases in MVPA over time

8. Secondary Outcome: Moderate-to-vigorous Physical Activity (Self-report)
Description: Change in physical activity from baseline to 3 months as measured using the Paffenbarger Physical Activity Questionnaire (PPAQ). The PPAQ assesses the amount of planned and lifestyle associated physical activity performed during a typical week. The PPAQ consists of three components: (1) stair climbing, (2) walking, and (3) sports and recreation. Participants report the frequency and duration of physical activity in the past week. PA Activities were classified as light, moderate, and vigorous based on their metabolic equivalent (MET) value and commonly used cut points. Moderate and vigorous activities were combined for self-reported minutes per week of MVPA. Range is 0 - no theoretical maximum.
Time Frame: Baseline, 3 months.
Population: ITT: all randomized participants using all PPAQ data.
Measure: Mean (95% Confidence Interval); unit: min/wk
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly)
Number analyzed (Participants) | 34 | 38 | 34 | 38 | 36 | 36 | 34 | 38
min/wk | 55.60 [3.13 to 108.07] | 34.13 [-17.03 to 85.29] | 50.97 [-4.77 to 106.71] | 38.76 [-9.53 to 87.05] | 47.36 [-3.83 to 98.55] | 42.37 [-10.18 to 94.92] | 58.67 [5.67 to 111.68] | 31.06 [-19.70 to 81.81]
Statistical Analysis 1: Comparison: Simplified Dietary Monitoring (Green) vs Simplified Dietary Monitoring (Red) vs Nutrition Goals (Yes) vs Nutrition Goals (No) vs Supportive Text Messages (Yes) vs Supportive Text Messages (No) vs Lesson Delivery (Once) vs Lesson Delivery (Weekly); Test type: Superiority — ITT analysis using linear mixed models comparing self-reported MVPA change over time (from baseline to 3 months). We fit a linear mixed model that included a random effect for participant and predictors (fixed effects) included time (baseline vs. follow-up) and all 4 factors; p = 0.004, Mixed Models Analysis; DF(2,127); Mean Difference (Net) = 44.87, 95% CI 2-sided [14.39 to 75.43] — The positive parameter estimate indicates an increase in self-reported MVPA over time for the full sample
Statistical Analysis 2: Comparison: Simplified Dietary Monitoring (Green) vs Simplified Dietary Monitoring (Red); ITT analysis for factor 1 (dietary self-monitoring) using linear mixed models comparing the effect of simplified dietary monitoring (green vs. red) on self-reported MVPA change over time (from baseline to 3 months); Test type: Superiority; p = 0.47, Mixed Models Analysis; DF(1,72); Mean Difference (Net) = -15.32, 95% CI 2-sided [-58.96 to 28.32] — Green food monitoring (reference) vs red food monitoring; a negative estimation parameter indicates that the non-referent group had greater increases in MVPA over time
Statistical Analysis 3: Comparison: Nutrition Goals (Yes) vs Nutrition Goals (No); ITT analysis for factor 2 (dietary goals) using linear mixed models comparing the effect of dietary goals (yes vs. no) on self-reported MVPA change over time (from baseline to 3 months); Test type: Superiority; p = 0.47, Mixed Models Analysis; DF(1,73); Mean Difference (Net) = 16.02, 95% CI 2-sided [-27.67 to 59.7] — Nutrition goals (yes; reference) vs no goals provided; a positive estimation parameter indicates that the reference group had greater increases in self-reported MVPA over time
Statistical Analysis 4: Comparison: Supportive Text Messages (Yes) vs Supportive Text Messages (No); ITT analysis for factor 3 (supportive text messages) using linear mixed models comparing the effect of text messages (yes vs. no) on self-reported MVPA change over time (from baseline to 3 months); Test type: Superiority; p = 0.66, Mixed Models Analysis; DF(1,71); Mean Difference (Net) = 9.72, 95% CI 2-sided [-34.09 to 53.52] — Supportive text messages (yes; reference) vs no text messages; a positive estimation parameter indicates that the reference group had greater increases in self-reported MVPA over time
Statistical Analysis 5: Comparison: Lesson Delivery (Once) vs Lesson Delivery (Weekly); ITT analysis for factor 4 (lesson delivery) using linear mixed models comparing the effect of lesson timing (once vs. weekly) on self-reported MVPA change over time (from baseline to 3 months); Test type: Superiority; p = 0.06, Mixed Models Analysis; DF(1,72); Mean Difference (Net) = -42.15, 95% CI 2-sided [-86.04 to 1.73] — Lesson delivery once (reference) vs weekly; a negative estimation parameter indicates that the non-referent group had greater increases in self-reported MVPA over time

9. Secondary Outcome: Dietary Intake: Healthy Eating Index (HEI)
Description: Dietary intake will be defined as the change in HEI score as measured by the NCI's Automated Self-Administered 24-hour (ASA 24-hour) dietary recalls from baseline to 3 months.The HEI consists of 13 component scores, including: total fruit, whole fruit, total protein foods, total vegetables, greens and beans, whole grains, dairy, seafood and plant proteins, fatty acids, sodium, refined grains, added sugars, and saturated fats. The summation of the 13 component scores ranges from 0 to 100, with higher scores indicating closer compliance with the Dietary Guidelines for Americans. Estimated mean change in HEI from baseline to 3 months for each of the two levels of each component obtained from intent-to-treat (ITT) linear mixed models of analysis of variance.
Time Frame: Baseline, 3 months
Population: ITT: all randomized participants using all available ASA24 data.
Measure: Mean (99% Confidence Interval); unit: Points
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly)
Number analyzed (Participants) | 34 | 38 | 34 | 38 | 36 | 36 | 34 | 38
Points | 4.66 [0.29 to 9.02] | 0.32 [-4.01 to 4.64] | 4.65 [-0.05 to 9.35] | 0.32 [-3.69 to 4.34] | 1.85 [-2.39 to 6.09] | 3.13 [-1.36 to 7.61] | 3.38 [-1.04 to 7.80] | 1.59 [-2.71 to 5.90]
Statistical Analysis 1: Comparison: Simplified Dietary Monitoring (Green) vs Simplified Dietary Monitoring (Red) vs Nutrition Goals (Yes) vs Nutrition Goals (No) vs Supportive Text Messages (Yes) vs Supportive Text Messages (No) vs Lesson Delivery (Once) vs Lesson Delivery (Weekly); ITT analysis using linear mixed models comparing HEI score change over time (from baseline to 3 months). We fit a linear mixed model that included a random effect for participant and predictors (fixed effects) included time (baseline vs. follow-up) and all 4 factors; Test type: Superiority; p = 0.109, Mixed Models Analysis; DF(1,61); Mean Difference (Net) = 2.49, 95% CI 2-sided [-0.56 to 5.54] — The positive parameter estimate indicates an increase in HEI score over time for the full sample
Statistical Analysis 2: Comparison: Simplified Dietary Monitoring (Green) vs Simplified Dietary Monitoring (Red); ITT analysis for factor 1 (dietary self-monitoring) using linear mixed models comparing the effect of simplified dietary monitoring (green vs. red) on HEI score change over time (from baseline to 3 months); Test type: Superiority; p = 0.71, Mixed Models Analysis; DF(1,68); Mean Difference (Net) = -1.17, 95% CI 2-sided [-7.42 to 5.08] — Green food monitoring (reference) vs red food monitoring; a negative estimation parameter indicates that the non-referent group had greater increases in HEI score
Statistical Analysis 3: Comparison: Nutrition Goals (Yes) vs Nutrition Goals (No); ITT analysis for factor 2 (dietary goals) using linear mixed models comparing the effect of dietary goals (yes vs. no) on HEI score change over time (from baseline to 3 months); Test type: Superiority; p = 0.89, Mixed Models Analysis; DF(1,68); Mean Difference (Net) = 0.44, 95% CI 2-sided [-5.82 to 6.69] — Nutrition goals (yes; reference) vs no goals provided; a positive estimation parameter indicates that the reference group had greater increases in HEI score over time
Statistical Analysis 4: Comparison: Supportive Text Messages (Yes) vs Supportive Text Messages (No); ITT analysis for factor 3 (supportive text messages) using linear mixed models comparing the effect of text messages (yes vs. no) on HEI score change over time (from baseline to 3 months); Test type: Superiority; p = 0.25, Mixed Models Analysis; DF(1,68); Mean Difference (Net) = 3.66, 95% CI 2-sided [-2.61 to 9.93] — Supportive text messages (yes; reference) vs no text messages; a positive estimation parameter indicates that the reference group had greater increases in HEI score over time
Statistical Analysis 5: Comparison: Lesson Delivery (Once) vs Lesson Delivery (Weekly); ITT analysis for factor 4 (lesson delivery) using linear mixed models comparing the effect of lesson timing (once vs. weekly) on HEI score change over time (from baseline to 3 months); Test type: Superiority; p = 0.57, Mixed Models Analysis; DF(1,68); Mean Difference (Net) = -1.83, 95% CI 2-sided [-8.11 to 4.45] — Lesson delivery once (reference) vs weekly; a negative estimation parameter indicates that the non-referent group had greater increases in HEI score over time

10. Secondary Outcome: Weight (kg)
Description: Estimated mean weight change in kg from baseline to 3 months. More negative values of weight change indicate greater weight loss (3-month weight - baseline weight).
Time Frame: Baseline, 3 months
Population: ITT: all randomized participants using all available weights.
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly)
Number analyzed (Participants) | 34 | 38 | 34 | 38 | 36 | 36 | 34 | 38
pounds | -1.47 [-3.44 to 0.51] | -2.39 [-4.38 to -0.40] | -1.26 [-3.40 to 0.87] | -2.60 [-4.43 to -0.76] | -2.32 [-4.27 to -0.36] | -1.54 [-3.56 to 0.48] | -2.23 [-4.28 to -0.18] | -1.63 [-3.55 to 0.29]

11. Secondary Outcome: Fried Physical Frailty : FRAIL Index
Description: The FRAIL Questionnaire includes five components that assess: 1) self-reported fatigue (PROMIS Fatigue Short form), 2) weight loss, 3) comorbidities (11 items from University of North Carolina Health Registry Comorbidity Assessment), 4) difficulty with ambulation (1 item from PROMIS Physical Function Short Form), and 5) ability to overcome resistance (1 item from PROMIS Physical Function)). The number of positive responses for these components is summed to create the FRAIL index (range 0-5) and characterized as "Frailty Status"; 0-1: robust, 2: prefrail, and 3+: frail. Changes in Frailty Status from baseline to 3 months will be assessed.
Time Frame: Baseline, 3 Months
Population: All randomized were characterized by Frailty Status (Robust, Prefrail, Frail) at baseline and 3-months. At 3 months, NA = insufficient data for classification based on missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly)
Number analyzed (Participants) | 34 | 38 | 34 | 38 | 36 | 36 | 34 | 38
Participants
  Baseline Frailty Status: Robust | 34 | 34 | 32 | 36 | 35 | 33 | 32 | 36
  Baseline Frailty Status: Prefrail | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
  Baseline Frailty Status: Frail | 0 | 3 | 2 | 1 | 1 | 2 | 2 | 1
  Baseline Frailty Status: NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  3-Month Frailty Status: Robust | 29 | 25 | 22 | 32 | 27 | 27 | 27 | 27
  3-Month Frailty Status: Prefrail | 1 | 6 | 2 | 5 | 5 | 2 | 3 | 4
  3-Month Frailty Status: Frail | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  3-Month Frailty Status: NA | 4 | 7 | 10 | 1 | 4 | 7 | 4 | 7

12. Secondary Outcome: Health-related Quality of Life: AYA PROMIS PRO Core Battery
Description: Changes in health-related quality of life from baseline to 3 months as measured using the Adolescent and Young Adult (AYA) PROMIS PRO Core Battery. These measures assess relevant HRQoL domains for AYA cancer survivors that are most likely to be impacted during and after cancer treatment. The AYA PRO Core battery includes the following PROMIS short forms: depression, anxiety, fatigue, physical function, pain interference, emotional support, and cognitive function. For each measure, each question has five responses ranging in value from 1 to 5, which are summed to find the total raw score. Total raw scores are translated to a T-score, standardized with a population mean of 50 and a standard deviation of 10. A higher PROMIS T-score represents more of the concept being measured.
Time Frame: Baseline, 3 months
Population: Participants who completed the PROMIS measures at 3 months.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- All Participants: All randomized participants
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly) | All Participants
Number analyzed (Participants) | 30 | 31 | 24 | 37 | 32 | 29 | 30 | 31 | 61
T-score
  Depressive Symptoms (PROMIS v1.0-Depression Short Form 4a) | 1.68 (9.19) | -1.85 (5.83) | 1.72 (9.87) | -1.3 (5.97) | 1.75 (9.01) | -2.17 (5.68) | -1.70 (7.71) | 1.42 (7.71) | -0.11 (7.81)
  Anxiety (PROMIS v1.0-Emotional Distress Anxiety Short Form 4a) | -1.50 (7.53) | -1.14 (7.95) | -0.83 (9.24) | -1.63 (6.51) | -1.76 (6.28) | -0.83 (9.07) | -1.41 (8.89) | -1.23 (6.45) | -1.32 (7.68)
  Fatigue (PROMIS v1.0-Fatigue Short form 4a) | -4.26 (9.64) | -0.65 (9.08) | -3.28 (7.34) | -1.87 (10.7) | -3.45 (9.67) | -1.29 (9.26) | -2.64 (10.8) | -2.22 (8.14) | -2.42 (9.46)
  Physical Function (PROMIS v2.0 Physical Function Short Form 4a) | 1.08 (5.29) | 0.60 (6.79) | -0.86 (6.28) | 1.94 (5.71) | 0.25 (4.78) | 1.49 (7.23) | 1.55 (5.14) | 0.15 (6.83) | 0.84 (6.05)
  Pain Interference (PROMIS v1.1 Pain Interference Short Form 4a) | 3.37 (6.12) | 2.65 (6.19) | 3.30 (5.45) | 2.81 (6.57) | 3.16 (6.61) | 2.83 (5.62) | 1.85 (4.92) | 4.12 (6.98) | 3.00 (6.11)
  Emotional Support (PROMIS v2.0 Emotional Support Short Form 4a) | -2.06 (6.22) | -0.003 (5.57) | -1.33 (6.05) | -0.81 (5.94) | -2.42 (6.67) | 0.54 (4.64) | -0.08 (5.90) | -1.91 (5.93) | -1.01 (5.94)
  Cognitive Function (PROMIS v2.0 Cognitive Function Short Form 4a) | 2.86 (8.67) | 1.48 (6.30) | 3.30 (7.56) | 1.41 (7.51) | 1.18 (7.10) | 3.24 (7.95) | 2.81 (9.03) | 1.53 (5.79) | 2.16 (7.52)

13. Secondary Outcome: Health-related Quality of Life: AYA PROMIS PRO Core Battery (Pain Intensity)
Description: Changes in health-related quality of life from baseline to 3 months as measured using the Adolescent and Young Adult (AYA) PROMIS PRO Core Battery. Pain intensity was assessed with the 1-tiem PROMIS v1.0 pain intensity 1a, "In the past 7 days, how would you rate your pain on average?" Scored 0-10 from no pain to the worst imaginable pain.
Time Frame: Baseline, 3 months
Population: Participants who completed the PROMIS measures at 3 months.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly) | All Participants
Number analyzed (Participants) | 30 | 31 | 24 | 37 | 32 | 29 | 30 | 31 | 61
Score on scale | 0.7 (2.12) | 0.36 (1.33) | 0.54 (1.47) | 0.51 (1.94) | 0.44 (1.54) | 0.62 (1.99) | 0.37 (1.81) | 0.68 (1.72) | 0.53 (1.76)

14. Secondary Outcome: Competence for Exercise and Nutrition
Description: Changes in perceived competence from baseline to 3 months as measured using the Perceived Competence Scale. The Scale measures perceived competence for diet (4 items) and physical activity (4 items). Items are rated on a 7-point Likert scale (1 = not at all true, 7 = very true), and include items such as "I feel confident in my ability to maintain a healthy diet." Scores are summed for the items in the subscale (diet and physical activity) and the range for each subscale is 4 - 28. Greater values indicate higher levels of perceived competence for engaging in positive diet and physical activity behaviors. Scores are summed for the items in each subscale separately (diet and physical activity). Outcomes are change in perceived competence for diet and change in perceived competence.
Time Frame: Baseline, 3 months
Population: Participants who completed the Perceived Competence Scales for Nutrition and Diet at 3 months
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly) | All Participants
Number analyzed (Participants) | 30 | 31 | 24 | 37 | 32 | 29 | 30 | 31 | 61
Score on scale
  Perceived Competence for Exercise | 0.6 (6.15) | -1.61 (4.09) | -1.38 (5.52) | 0.027 (5.12) | -1.28 (5.13) | 0.31 (5.41) | 0.9 (5.51) | -1.90 (4.74) | -0.53 (5.28)
  Perceived Competence for Nutrition | 1.13 (4.49) | -0.03 (2.98) | 0.54 (4.53) | 0.54 (3.34) | 0.28 (4.11) | 0.83 (3.51) | 1.53 (3.14) | -0.42 (4.20) | 0.54 (3.81)

15. Secondary Outcome: Self-efficacy for Exercise and Nutrition
Description: Changes in self-efficacy from baseline to 3 months as measured using the Nutrition and Physical Activity Self-Efficacy Scale, a 10-items measured on a 4-point Likert scale that assesses an individual's confidence (where where 1 is 'very uncertain' to 4 'very certain') with in their ability to eat healthy foods (5 items) and exercise (5 items) in the presence of barriers. Self-efficacy for each behavior is calculated as the sum of the 5 Likert-type responses with a range of 5-20 for each subscale. Higher values indicate higher levels of self-efficacy for the behavior. Outcomes are changes in self-eficacy for exercise and self-efficacy for nutrition from baseline to 3 months.
Time Frame: Baseline, 3 months
Population: Participants who completed the Self-efficacy Scale for Exercise and Diet at 3 months.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly) | All Participants
Number analyzed (Participants) | 30 | 31 | 24 | 37 | 32 | 29 | 30 | 31 | 61
Score on scale
  Self-efficacy for Exercise | -0.3 (3.80) | 0.06 (2.46) | 0.58 (3.71) | -0.57 (2.72) | 0 (3.34) | -0.24 (3.02) | -0.27 (2.72) | 0.03 (3.59) | -0.12 (3.17)
  Self-efficacy for Nutrition | 0.73 (2.94) | 0.39 (2.53) | 0.71 (2.74) | 0.46 (2.73) | 1.25 (2.83) | -0.21 (2.41) | 0.53 (2.43) | 0.58 (3.01) | 0.56 (2.72)

16. Secondary Outcome: Self-Regulation for Exercise and Nutrition
Description: Changes in self-regulation from baseline to 3 months as measured using the Treatment Self-Regulation Questionnaire (TSRQ). The TSRQ assesses autonomous and controlled motivation for making changes in diet (15 items) and physical activity (15 items). Ratings are on a 7-point Likert scale indicating agreement with statements regarding motivation for behavior change. Examples item: "Because I feel that I want to take responsibility for my own health" answered on a scale of 1 (not at all true) to 7 (very true)." Calculating the scores for the sub-scales will consist of averaging the items on that subscale. Responses to the items within the subscale are averaged with the range of scores being 1 to 7. Higher values on each subscale indicate greater levels of that type of motivation. Outcomes are changes in autonomous and controlled motivation for exercise and diet at 3 months.
Time Frame: Baseline, 3 months
Population: Participants who completed the Treatment Self-Regulation Questionnaire (TSRQ) for Exercise and Diet at 3 months.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly) | All Participants
Number analyzed (Participants) | 30 | 31 | 24 | 37 | 32 | 29 | 30 | 31 | 61
Score on scale
  Autonomous Motivation for Exercise | -0.06 (0.85) | -0.09 (0.761) | -0.17 (0.87) | -0.014 (0.76) | 0.04 (0.88) | -0.20 (0.70) | -0.04 (0.76) | -0.11 (0.85) | -0.07 (0.80)
  Autonomous Motivation for Diet | -0.07 (0.88) | 0.02 (0.71) | -0.11 (0.89) | 0.04 (0.74) | -0.05 (1.01) | 0.006 (0.48) | -0.03 (0.53) | -0.02 (1.0) | -0.02 (0.80)
  Externally Controlled Motivation for Exercise | -0.01 (0.61) | 0.38 (1.05) | 0.05 (1.04) | 0.28 (0.76) | 0.14 (0.95) | 0.24 (0.81) | 0.44 (0.82) | -0.07 (0.88) | 0.19 (0.88)
  Externally Controlled Motivation for Diet | 0 (0.96) | 0.27 (0.95) | -0.13 (0.89) | 0.31 (0.97) | 0.03 (1.12) | 0.26 (0.73) | 0.12 (0.80) | 0.15 (1.10) | 0.14 (0.96)

17. Secondary Outcome: Autonomy Support
Description: Changes in perceived autonomy support from baseline to 3 months as measured using the Virtual Care Climate Questionnaire (VCCQ) a 15-item measure of perceived support for autonomy provided by the study team in a virtual care setting. Ratings are on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). Responses are averaged with a range of 1 to 7. Higher scores indicate a higher level of perceived autonomy support in a virtual setting.
Time Frame: Baseline, 3 months
Population: Participants who completed the Virtual Care Climate Questionnaire (VCCQ) at 3 months.
Measure: Median (Standard Deviation); unit: Score on scale
Arm/Group | Simplified Dietary Monitoring (Green) | Simplified Dietary Monitoring (Red) | Nutrition Goals (Yes) | Nutrition Goals (No) | Supportive Text Messages (Yes) | Supportive Text Messages (No) | Lesson Delivery (Once) | Lesson Delivery (Weekly) | All Participants
Number analyzed (Participants) | 30 | 30 | 24 | 36 | 31 | 29 | 30 | 30 | 60
Score on scale | 4.98 (1.06) | 4.84 (1.13) | 4.59 (0.89) | 5.12 (1.16) | 4.97 (1.24) | 4.85 (0.92) | 5.07 (1.18) | 4.75 (0.98) | 4.91 (1.09)

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/4 | 0/4 | 0/3 | 0/4 | 0/6 | 0/4 | 0/2 | 0/5 | 0/5 | 0/5 | 0/6 | 0/7 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 1/4 | 0/4 | 0/3 | 0/4 | 0/6 | 0/4 | 0/2 | 0/5 | 0/5 | 0/5 | 0/6 | 0/7 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 4/5 | 0/4 | 3/4 | 2/3 | 1/4 | 1/6 | 2/4 | 1/2 | 3/5 | 3/5 | 3/5 | 3/6 | 4/7 | 1/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Condition 1 (N=4) | Condition 2 (N=5) | Condition 3 (N=4) | Condition 4 (N=4) | Condition 5 (N=3) | Condition 6 (N=4) | Condition 7 (N=6) | Condition 8 (N=4) | Condition 9 (N=2) | Condition 10 (N=5) | Condition 11 (N=5) | Condition 12 (N=5) | Condition 13 (N=6) | Condition 14 (N=7) | Condition 15 (N=4) | Condition 16 (N=4)
Bowel Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Hospitalized for 2 nights
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Condition 1 (N=4) | Condition 2 (N=5) | Condition 3 (N=4) | Condition 4 (N=4) | Condition 5 (N=3) | Condition 6 (N=4) | Condition 7 (N=6) | Condition 8 (N=4) | Condition 9 (N=2) | Condition 10 (N=5) | Condition 11 (N=5) | Condition 12 (N=5) | Condition 13 (N=6) | Condition 14 (N=7) | Condition 15 (N=4) | Condition 16 (N=4)
Racing heartbeat (Cardiac disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Resolved <24 hrs, no other detail provided
Low blood pressure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PVCs (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Motor vehicle accident (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throbbing back and hip pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Related to motor vehicle accident
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis in shoulder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress injury in tibia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bruised/cracked rib from bronchitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0
Headaches and neck pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Pulled out lower back, neck, and shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Due to walking around for an extended period of time at a music festival
Lymphadema flare (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Debilitating menstrual cramps (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Tweaked IT band (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Not related to intervention
Migraine (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Bruised hip (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Twisted ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus infection/sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid, cold, flu, viral illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2) — Impacted ability to exercise

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT05887401/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT05887401/ICF_001.pdf